CLINICAL TRIAL: NCT04156360
Title: Construction and Evaluation of the Liquid Biopsy-based Early Diagnostic Model for Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Director Head of Medical Oncology, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: YT2019-001
Record Dates: First submitted 2019-10-28; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Healthy; Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers
- Patients With Pulmonary Nodule

SUMMARY:
The purpose of this study is to detetct Circulating tumor cells(CTCs) and Cancer Associated Macrophage-Like cells (CAMLs) in patients with pulmonary nodules using a novel microfluidic CTC-detection system. Then construct an early diagnostic model for lung cancer.

DETAILED DESCRIPTION:
Patients found pulmonary nodules by CT screening will be enrolled in this study prospectively. CTCs and CAMLs both are cancer specific biomarkers found in the peripheral blood of patients with solid tumors including lung cancer. Through detecting CTCs and CAMLs in healthy volunteers and patients with pulmonary nodules who undergo biopsy, determine the cut-off value of the test. Further analysis of the test specificity and sensitivity, and on this basis construct an early diagnostic model for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18 years of age or older
* Pulmonary nodules diagnosed by chest CT or low-dose computed tomography (LDCT) scans

Exclusion Criteria:

* Prior diagnosis of lung cancer or other invasive malignancy within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with pulmonary nodules diagnosed by chest CT or low-dose computed tomography (LDCT) scans
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Determination of prevalence of CTCs and CAMLs in patients with pulmonary nodules | 12 months
  The number of CTCs and CAMLs will be detected in the peripheral blood of patients with pulmonary nodules using a novel microfluidic CTC-detection system.

SECONDARY OUTCOMES:
Determination of optimal cut-off values for screening Lung Cancer paitents | 6 months
  The optimal cut-off values will be determined by the ROC analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Yayi He, MD, PHD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University